CLINICAL TRIAL: NCT05978999
Title: Blood Pressure Monitor#Model#BPM1#Clinical Test
Brief Title: Blood Pressure Monitor Clinical Test (Cuff Range: 15cm-24cm, 20cm-34cm, 30cm-44cm, 22cm-42cm)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Andon Health 12
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2022-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject use both BPM1 Arm Automatic Electronic BPM and mercury sphygmomanometers

SUMMARY:
The purpose of this study is to verify the accuracy of the 4 blood pressure cuffs with blood pressure monitor device.

Cuff circumference is : 15cm-24cm, 20cm-34cm, 30cm-44cm, 22cm-42cm

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure and hypertensive patients over 12 years old

Exclusion Criteria:

* Patients with serious arrhythmias or a high frequency of arrhythmias
* Pregnant woman
* Other investigators believe that it is not suitable to participate in this clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal blood pressure and hypertensive patients over 12 years old
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
blood pressure monitor accuracy | 30 minutes
  All the test results of the electronic blood pressure monitor with 4 cuffs is within the accuracy creteria, with the merury sphygmomanometer as control

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, China